CLINICAL TRIAL: NCT00444457
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of Three Lots of 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in the United States
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine In Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6096A1-3005
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Results first posted 2010-07-14 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Vaccines, Pneumococcal
Keywords: Vaccine; Infants; Pneumococcal Conjugate Vaccines; Vaccines, Pneumococcal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- 2 (Experimental)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- 3 (Experimental)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- 4 (Active Comparator)
  Interventions: Biological: 7vPnC

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — 0.5 mL of study vaccine administered IM at 2, 4, 6, and 12 months of age.
  Arms: 1; 2; 3
Biological: 7vPnC — 0.5 mL of study vaccine administered IM at 2, 4, 6, and 12 months of age.
  Arms: 4

SUMMARY:
The purpose of this study will be to evaluate safety, tolerability and immunogenicity of three lots of 13-valent pneumococcal vaccine given to healthy infants. Lots will be studied for consistency of the immune response, as well as for non-inferiority and safety as compared to 7-valent Pneumococcal Conjugate Vaccine.

ELIGIBILITY:
Inclusion criteria:

* Healthy 2 month old infants
* Available for the duration of the study and reachable by telephone
* Able to complete two blood drawing procedures during the study

Exclusion criteria:

* Previous vaccination, contraindication or history of allergic reaction to vaccines or vaccine components
* Bleeding disorder, immune deficiency or significant chronic or congenital disease
* Previous receipt of blood products or immune globulin

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1712 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (70):
- United States (70):
  - Benton, Arkansas
  - Conway, Arkansas
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Downey, California
  - Fontana, California
  - Fountain Valley, California
  - Lakewood, California
  - Loma Linda, California
  - Moreno Valley, California
  - Paramount, California
  - Riverside, California
  - Rolling Hills Estates, California
  - Boulder, Colorado
  - Longmont, Colorado
  - Norwich, Connecticut
  - Palm Beach Gardens, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Woodstock, Georgia
  - Nampa, Idaho
  - Chicago, Illinois
  - DeKalb, Illinois
  - Bardstown, Kentucky
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Jamaica Plain, Massachusetts
  - Jackson, Mississippi
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Whitehouse Station, New Jersey
  - Fishkill, New York
  - Hopewell Jct, New York
  - Ithaca, New York
  - Syracuse, New York
  - The Bronx, New York
  - Cary, North Carolina
  - Durham, North Carolina
  - Sylva, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Huber Heights, Ohio
  - Kettering, Ohio
  - Mason, Ohio
  - Tulsa, Oklahoma
  - Kittanning, Pennsylvania
  - Latrobe, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Clarksville, Tennessee
  - Franklin, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Galveston, Texas
  - San Antonio, Texas
  - Layton, Utah
  - Murray, Utah
  - South Jordan, Utah
  - Vienna, Virginia
  - Vancouver, Washington
  - La Crosse, Wisconsin
  - Marshfield, Wisconsin
  - Monroe, Wisconsin

REFERENCES:
- [Derived] Payton T, Girgenti D, Frenck RW, Patterson S, Love J, Razmpour A, Sidhu MS, Emini EA, Gruber WC, Scott DA. Immunogenicity, safety and tolerability of 3 lots of 13-valent pneumococcal conjugate vaccine given with routine pediatric vaccinations in the United States. Pediatr Infect Dis J. 2013 Aug;32(8):871-80. doi: 10.1097/INF.0b013e3182906499. PMID 23584582
- [Derived] Bryant KA, Gurtman A, Girgenti D, Reisinger K, Johnson A, Pride MW, Patterson S, Devlin C, Gruber WC, Emini EA, Scott DA. Antibody responses to routine pediatric vaccines administered with 13-valent pneumococcal conjugate vaccine. Pediatr Infect Dis J. 2013 Apr;32(4):383-8. doi: 10.1097/INF.0b013e318279e9a9. PMID 23104129

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC (Pilot Lot 1): Participants received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 1 at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age; a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age.
- 13vPnC (Pilot Lot 2): Participants received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 2 at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age; a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age.
- 13vPnC (Manufacturing Lot): Participants received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) manufacturing lot (manu lot) at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age; a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age.
- 7vPnC: Participants received 1 single 0.5 milliliter (mL) dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age; a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age.
Period: Infant Series
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Started | 489 | 488 | 489 | 246
Vaccinated Dose 1 | 486 | 484 | 485 | 244
Vaccinated Dose 2 | 455 | 447 | 455 | 228
Vaccinated Dose 3 | 442 | 435 | 438 | 225
Completed | 435 | 427 | 428 | 218
Not Completed | 54 | 61 | 61 | 28
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Parent or legal guardian request | 18 | 29 | 34 | 14
Not completed — Lost to Follow-up | 10 | 11 | 7 | 6
Not completed — Protocol Violation | 16 | 8 | 6 | 3
Not completed — Failed to return | 5 | 4 | 4 | 2
Not completed — Investigator request | 4 | 3 | 3 | 2
Not completed — Other | 0 | 2 | 4 | 0
Not completed — Adverse Event | 1 | 2 | 2 | 0
Not completed — Death | 0 | 1 | 1 | 1
Period: After Infant Series
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Started | 435 | 427 | 427 | 218
Completed | 415 (Not completed=Withdrawn after infant series) | 397 (Not completed=Withdrawn after infant series) | 408 (Not completed=Withdrawn after infant series) | 208 (Not completed=Withdrawn after infant series)
Not Completed | 20 | 30 | 19 | 10
Not completed — Other | 0 | 1 | 1 | 1
Not completed — Parent or legal guardian request | 4 | 11 | 6 | 3
Not completed — Failed to return | 7 | 6 | 5 | 1
Not completed — Lost to Follow-up | 5 | 5 | 5 | 2
Not completed — Protocol Violation | 2 | 4 | 2 | 2
Not completed — Adverse Event | 2 | 2 | 0 | 0
Not completed — Investigator request | 0 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0
Period: Toddler Dose
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Started | 415 (Vaccinated toddler dose) | 397 (Vaccinated toddler dose) | 408 (Vaccinated toddler dose) | 208 (Vaccinated toddler dose)
Completed | 408 | 391 | 404 | 200
Not Completed | 7 | 6 | 4 | 8
Not completed — Lost to Follow-up | 4 | 1 | 1 | 3
Not completed — Failed to return | 2 | 2 | 1 | 3
Not completed — Parent or legal guardian request | 0 | 3 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC | Total
Number analyzed (Participants) | 489 | 488 | 489 | 246 | 1712
Age Continuous [Mean (Standard Deviation); unit: months] | 2.2 (0.3) | 2.2 (0.3) | 2.2 (0.3) | 2.2 (0.3) | 2.2 (0.3)
Sex/Gender, Customized [Number; unit: participants]
  Female | 230 | 226 | 213 | 115 | 784
  Male | 259 | 260 | 275 | 131 | 925
  Unknown | 0 | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody in the Three 13vPnC Groups 1 Month After the Infant Series
Description: Antibody geometric mean concentration (GMC) as measured by micrograms per milliliter (mcg/mL) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 Month after the infant series (7 Months of age)
Population: Evaluable immunogenicity population: treatments as randomized at all expected doses, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations; (n)=number of participants with IgG antibody concentration to given serotype for the three 13vPnC lots, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: GMC mcg/mL
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot)
Number analyzed (Participants) | 435 | 427 | 427
GMC mcg/mL
  Common serotypes - serotype 4 (n=411, 404, 398) | 1.33 [1.24 to 1.43] | 1.34 [1.25 to 1.44] | 1.75 [1.63 to 1.88]
  Common serotypes - serotype 6B (n=409, 401, 396) | 2.89 [2.58 to 3.23] | 2.15 [1.91 to 2.42] | 2.54 [2.27 to 2.85]
  Common serotypes - serotype 9V (n=411, 403, 396) | 1.05 [0.98 to 1.12] | 1.11 [1.04 to 1.19] | 1.11 [1.04 to 1.19]
  Common serotypes - serotype 14 (n=398. 387, 387) | 4.97 [4.59 to 5.37] | 5.13 [4.70 to 5.59] | 5.18 [4.72 to 5.69]
  Common serotypes - serotype 18C (n=413, 401, 398) | 1.30 [1.22 to 1.38] | 1.34 [1.24 to 1.44] | 1.48 [1.38 to 1.58]
  Common serotypes - serotype 19F (n=408, 399, 398) | 1.85 [1.71 to 1.99] | 2.07 [1.92 to 2.24] | 2.59 [2.40 to 2.78]
  Common serotypes - serotype 23F (n=411, 402, 399) | 1.24 [1.13 to 1.36] | 1.27 [1.15 to 1.40] | 1.03 [0.94 to 1.14]
  Additional serotypes - serotype 1 (n=411, 403,395) | 1.62 [1.50 to 1.76] | 1.81 [1.66 to 1.98] | 1.91 [1.76 to 2.07]
  Additional serotypes - serotype 3 (n=406, 391,393) | 0.52 [0.48 to 0.55] | 0.56 [0.52 to 0.61] | 0.61 [0.57 to 0.66]
  Additional serotypes - serotype 5 (n=412, 402,393) | 1.35 [1.24 to 1.47] | 1.05 [0.96 to 1.14] | 1.35 [1.25 to 1.47]
  Additional serotypes - serotype 6A (n=413,402,398) | 2.40 [2.21 to 2.61] | 2.10 [1.92 to 2.29] | 2.12 [1.96 to 2.30]
  Additional serotypes - serotype 7F (n=412,401,397) | 2.54 [2.37 to 2.71] | 2.52 [2.35 to 2.70] | 2.67 [2.50 to 2.85]
  Additional serotype - serotype 19A (n=411,403,397) | 1.85 [1.71 to 2.00] | 2.00 [1.85 to 2.16] | 1.88 [1.74 to 2.02]
Statistical Analysis 1: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — The 3 lots were considered equivalent if the maximum difference between any 2 lots is less than 0.693 and greater than -0.693 using the equivalence testing procedure for 3 vaccine groups given by Wiens and Iglewicz, for all 13 serotypes; difference in log-transformed GM = -0.01, 95% CI 2-sided [-0.11 to 0.09] — 2-sided 95% CI were constructed by back transformation of the CI for the mean of the logarithmically transformed assay results computed using the Student t distribution
Statistical Analysis 2: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.27, 95% CI 2-sided [-0.38 to -0.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.27, 95% CI 2-sided [-0.37 to -0.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.30, 95% CI 2-sided [0.13 to 0.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.13, 95% CI 2-sided [-0.04 to 0.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.17, 95% CI 2-sided [-0.33 to -0.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.06, 95% CI 2-sided [-0.16 to 0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.06, 95% CI 2-sided [-0.16 to 0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.00, 95% CI 2-sided [-0.10 to 0.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.03, 95% CI 2-sided [-0.15 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.04, 95% CI 2-sided [-0.16 to 0.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.01, 95% CI 2-sided [-0.13 to 0.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.03, 95% CI 2-sided [-0.13 to 0.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.13, 95% CI 2-sided [-0.23 to -0.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.10, 95% CI 2-sided [-0.20 to -0.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.11, 95% CI 2-sided [-0.22 to -0.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.34, 95% CI 2-sided [-0.44 to -0.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.22, 95% CI 2-sided [-0.33 to -0.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.03, 95% CI 2-sided [-0.16 to 0.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.18, 95% CI 2-sided [0.04 to 0.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.20, 95% CI 2-sided [0.07 to 0.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.11, 95% CI 2-sided [-0.23 to 0.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.16, 95% CI 2-sided [-0.28 to -0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.05, 95% CI 2-sided [-0.17 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.09, 95% CI 2-sided [-0.19 to 0.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.18, 95% CI 2-sided [-0.28 to -0.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.09, 95% CI 2-sided [-0.19 to 0.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.25, 95% CI 2-sided [0.13 to 0.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 29: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.00, 95% CI 2-sided [-0.12 to 0.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 30: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.25, 95% CI 2-sided [-0.37 to -0.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 31: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.14, 95% CI 2-sided [0.02 to 0.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 32: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.12, 95% CI 2-sided [0.01 to 0.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 33: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.01, 95% CI 2-sided [-0.13 to 0.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 34: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.01, 95% CI 2-sided [-0.09 to 0.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 35: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.05, 95% CI 2-sided [-0.14 to 0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 36: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.06, 95% CI 2-sided [-0.15 to 0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 37: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.08, 95% CI 2-sided [-0.19 to 0.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 38: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = -0.02, 95% CI 2-sided [-0.12 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 39: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in log-transformed GM = 0.06, 95% CI 2-sided [-0.05 to 0.17] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Level ≥0.1 International Units Per Milliliter (IU/mL) for Tetanus Toxoid in the Combined 13vPnC Group Relative to 7vPnC Group 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥0.1 IU/ mL along with the corresponding 95% CI for concomitant antigen tetanus toxoid are presented. Exact 2-sided CI was based on the observed proportion of participants. Combined 13vPnC group includes participants randomized to pilot lot 1, pilot lot 2, or the manufacturing lot.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable immunogenicity population. Combined 13vPnC group includes participants who received pilot lot 1, pilot lot 2, or manufacturing lot; N=number of participants analyzed with a determinate post-third dose IgG antibody concentration to the given concomitant vaccine component.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Groups:
- Combined 13vPnC: Participants received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 1 or 2, or manufacturing lot at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age; a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age.
Arm/Group | Combined 13vPnC | 7vPnC
Number analyzed (Participants) | 184 | 196
observed percentage of participants | 98.4 [95.3 to 99.7] | 98.5 [95.6 to 99.7]
Statistical Analysis 1: Comparison: Combined 13vPnC vs 7vPnC; Tetanus toxoid: Difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — For each of the 5 concomitant antigens (tetanus toxoid, poliovirus Type 1, 2, and 3, and hepatitis b antibodies), non-inferiority was shown if the lower limit of the 2-sided 95% CI, computed using the Chan and Zhang procedure for the difference in proportions, is greater than -10%; Difference = -0.1, 95% CI 2-sided [-3.3 to 3.0] — Exact 2-sided CI for difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage

3. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Level ≥1:8 for Poliovirus in the Combined 13vPnC Group Relative to 7vPnC Group 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥1:8 along with the corresponding 95% CI for concomitant antigen poliovirus type 1, type 2, and type 3 (Sabin strains 1, 2, 3) are presented. Exact 2-sided CI was based on the observed proportion of participants. Combined 13vPnC group includes participants randomized to pilot lot 1, pilot lot 2, or the manufacturing lot.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable immunogenicity population; N=number of participants analyzed with a determinate post-third dose IgG antibody concentration to the given concomitant vaccine component; n)=number of participants with an antibody titer ≥ prespecified level for given concomitant vaccine antigen for combined 13vPnC and 7vPnC, respectively.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | Combined 13vPnC | 7vPnC
Number analyzed (Participants) | 183 | 187
observed percentage of participants
  Poliovirus type 1 (n=183, 187) | 100.0 [98.0 to 100.0] | 100.0 [98.0 to 100.0]
  Poliovirus type 2 (n=181, 186) | 98.9 [96.1 to 99.9] | 99.5 [97.1 to 100.0]
  Poliovirus type 3 (n=182, 186) | 100.0 [98.0 to 100.0] | 99.5 [97.1 to 100.0]
Statistical Analysis 1: Comparison: Combined 13vPnC vs 7vPnC; Poliovirus type 1: Difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference = 0.0, 95% CI 2-sided [-2.1 to 2.0] — Exact 2-sided CI for difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage
Statistical Analysis 2: Comparison: Combined 13vPnC vs 7vPnC; Poliovirus type 2: Difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference = -0.6, 95% CI 2-sided [-3.4 to 2.0] — Exact 2-sided CI for difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage
Statistical Analysis 3: Comparison: Combined 13vPnC vs 7vPnC; Poliovirus type 3: Difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference = 0.5, 95% CI 2-sided [-1.5 to 3.0] — Exact 2-sided CI for difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage

4. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Level ≥10.0 Milli-International Units Per Milliliter (mIU/mL) for Hepatitis B in the Combined 13vPnC Group Relative to 7vPnC Group 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥10.0 mIU/ mL along with the corresponding 95% CI for concomitant antigen hepatitis B are presented. Exact 2-sided CI was based on the observed proportion of participants. Combined 13vPnC group includes participants randomized to pilot lot 1, pilot lot 2, or the manufacturing lot.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable immunogenicity population; N=number of participants analyzed with a determinate post-third dose IgG antibody concentration to the given concomitant vaccine component.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | Combined 13vPnC | 7vPnC
Number analyzed (Participants) | 153 | 173
observed percentage of participants | 100.0 [97.6 to 100.0] | 100.0 [97.9 to 100.0]
Statistical Analysis 1: Comparison: Combined 13vPnC vs 7vPnC; Hepatitis B: Difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference = 0.0, 95% CI 2-sided [-2.4 to 2.2] — Exact 2-sided CI for difference in proportions (combined 13vPnC, 7vPnC) expressed as a percentage

5. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35 Mcg/mL in the Three 13vPnC Groups 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥0.35mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable immunogenicity population; (n)=number of subjects with a determinate IgG antibody concentration to the given serotype for the three 13vPnC lots, respectively.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot)
Number analyzed (Participants) | 435 | 427 | 427
observed percentage of participants
  Common serotypes - serotype 4 (n=411, 404, 398) | 97.6 [95.6 to 98.8] | 95.5 [93.0 to 97.3] | 98.5 [96.7 to 99.4]
  Common serotypes - serotype 6B (n=409, 401, 396) | 94.9 [92.3 to 96.8] | 89.5 [86.1 to 92.3] | 94.4 [91.7 to 96.5]
  Common serotypes - serotype 9V (n=411, 403, 396) | 95.4 [92.9 to 97.2] | 95.5 [93.0 to 97.3] | 96.5 [94.1 to 98.1]
  Common serotypes - serotype 14 (n=398, 387, 387) | 99.2 [97.8 to 99.8] | 99.0 [97.4 to 99.7] | 98.2 [96.3 to 99.3]
  Common serotypes - serotype 18C (n=413, 401, 398) | 97.8 [95.9 to 99.0] | 95.8 [93.3 to 97.5] | 98.0 [96.1 to 99.1]
  Common serotypes - serotype 19F (n=408, 399, 398) | 97.8 [95.9 to 99.0] | 97.5 [95.4 to 98.8] | 99.2 [97.8 to 99.8]
  Common serotypes - serotype 23F (n=411, 402, 399) | 91.2 [88.1 to 93.8] | 88.1 [84.5 to 91.1] | 87.2 [83.5 to 90.3]
  Additional serotypes - serotype 1 (n=411, 403,395) | 97.8 [95.9 to 99.0] | 97.0 [94.9 to 98.5] | 98.5 [96.7 to 99.4]
  Additional serotypes - serotype 3 (n=406, 391,393) | 68.5 [63.7 to 73.0] | 72.4 [67.7 to 76.8] | 79.1 [74.8 to 83.0]
  Additional serotypes - serotype 5 (n=412, 402,393) | 94.2 [91.5 to 96.2] | 90.3 [87.0 to 93.0] | 94.4 [91.6 to 96.5]
  Additional serotypes - serotype 6A (n=413,402,398) | 98.1 [96.2 to 99.2] | 95.5 [93.0 to 97.3] | 98.2 [96.4 to 99.3]
  Additional serotypes - serotype 7F (n=412,401,397) | 99.8 [98.7 to 100.0] | 99.0 [97.5 to 99.7] | 99.7 [98.6 to 100.0]
  Additional serotype - serotype 19A (n=411,403,397) | 98.1 [96.2 to 99.2] | 99.0 [97.5 to 99.7] | 98.7 [97.1 to 99.6]
Statistical Analysis 1: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — Exact, unconditional 2-sided 95% CI on the pairwise difference in proportions were computed using the noninferiority procedure of Chan and Zhang, using the standardized test statistics and gamma=0.000001; Difference = 2.0, 95% CI 2-sided [-0.51 to 4.75]
Statistical Analysis 2: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.9, 95% CI 2-sided [-3.09 to 1.10]
Statistical Analysis 3: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -2.9, 95% CI 2-sided [-5.58 to -0.58]
Statistical Analysis 4: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 5.3, 95% CI 2-sided [1.55 to 9.19]
Statistical Analysis 5: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.4, 95% CI 2-sided [-2.77 to 3.66]
Statistical Analysis 6: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -4.9, 95% CI 2-sided [-8.82 to -1.10]
Statistical Analysis 7: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.2, 95% CI 2-sided [-3.13 to 2.83]
Statistical Analysis 8: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -1.1, 95% CI 2-sided [-3.97 to 1.73]
Statistical Analysis 9: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.9, 95% CI 2-sided [-3.81 to 1.88]
Statistical Analysis 10: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.3, 95% CI 2-sided [-1.27 to 1.95]
Statistical Analysis 11: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 1.1, 95% CI 2-sided [-0.60 to 3.01]
Statistical Analysis 12: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.8, 95% CI 2-sided [-1.04 to 2.76]
Statistical Analysis 13: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 2.1, 95% CI 2-sided [-0.38 to 4.74]
Statistical Analysis 14: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.2, 95% CI 2-sided [-2.33 to 1.99]
Statistical Analysis 15: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -2.2, 95% CI 2-sided [-4.89 to 0.23]
Statistical Analysis 16: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.3, 95% CI 2-sided [-1.93 to 2.60]
Statistical Analysis 17: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -1.5, 95% CI 2-sided [-3.46 to 0.28]
Statistical Analysis 18: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -1.8, 95% CI 2-sided [-3.87 to 0.02]
Statistical Analysis 19: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 3.2, 95% CI 2-sided [-1.03 to 7.46]
Statistical Analysis 20: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 4.0, 95% CI 2-sided [-0.27 to 8.39]
Statistical Analysis 21: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.8, 95% CI 2-sided [-3.75 to 5.46]
Statistical Analysis 22: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.8, 95% CI 2-sided [-1.48 to 3.18]
Statistical Analysis 23: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.7, 95% CI 2-sided [-2.78 to 1.34]
Statistical Analysis 24: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -1.5, 95% CI 2-sided [-3.77 to 0.67]
Statistical Analysis 25: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -3.9, 95% CI 2-sided [-10.27 to 2.45]
Statistical Analysis 26: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -10.7, 95% CI 2-sided [-16.80 to -4.57]
Statistical Analysis 27: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -6.8, 95% CI 2-sided [-12.76 to -0.74]
Statistical Analysis 28: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 3.9, 95% CI 2-sided [0.15 to 7.69]
Statistical Analysis 29: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.2, 95% CI 2-sided [-3.52 to 3.09]
Statistical Analysis 30: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -4.1, 95% CI 2-sided [-7.92 to -0.36]
Statistical Analysis 31: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 2.5, 95% CI 2-sided [0.12 to 5.23]
Statistical Analysis 32: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.2, 95% CI 2-sided [-2.22 to 1.86]
Statistical Analysis 33: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -2.7, 95% CI 2-sided [-5.39 to -0.27]
Statistical Analysis 34: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.8, 95% CI 2-sided [-0.47 to 2.30]
Statistical Analysis 35: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.0, 95% CI 2-sided [-1.12 to 1.18]
Statistical Analysis 36: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.7, 95% CI 2-sided [-2.30 to 0.52]
Statistical Analysis 37: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -1.0, 95% CI 2-sided [-2.91 to 0.80]
Statistical Analysis 38: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = -0.7, 95% CI 2-sided [-2.69 to 1.19]
Statistical Analysis 39: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.3, 95% CI 2-sided [-1.40 to 2.04]

6. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35 Mcg/mL in the Three 13vPnC Groups 1 Month After the Toddler Dose
Description: Percentage of participants achieving predefined antibody threshold ≥0.35 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 month after the toddler dose (13 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot)
Number analyzed (Participants) | 415 | 397 | 408
observed percentage of participants
  Common serotypes - serotype 4 (n=364, 342, 355) | 99.2 [97.6 to 99.8] | 99.1 [97.5 to 99.8] | 100.0 [99.0 to 100.0]
  Common serotypes - serotype 6B (n=368,341,357) | 100.0 [99.0 to 100.0] | 100.0 [98.9 to 100.0] | 100.0 [99.0 to 100.0]
  Common serotypes - serotype 9V (n=368,342,357) | 99.7 [98.5 to 100.0] | 99.7 [98.4 to 100.0] | 99.2 [97.6 to 99.8]
  Common serotypes - serotype 14 (n=366,344,358) | 100.0 [99.0 to 100.0] | 99.7 [98.4 to 100.0] | 100.0 [99.0 to 100.0]
  Common serotypes - serotype 18C (n=362,341,354) | 98.9 [97.2 to 99.7] | 98.5 [96.6 to 99.5] | 99.4 [98.0 to 99.9]
  Common serotypes - serotype 19F (n=362,342,353) | 98.3 [96.4 to 99.4] | 98.8 [97.0 to 99.7] | 99.4 [98.0 to 99.9]
  Common serotypes - serotype 23F (n=362,340,353) | 99.4 [98.0 to 99.9] | 99.1 [97.4 to 99.8] | 98.3 [96.3 to 99.4]
  Additional serotypes - serotype 1 (n=367,344,357) | 100.0 [99.0 to 100.0] | 99.1 [97.5 to 99.8] | 99.2 [97.6 to 99.8]
  Additional serotypes - serotype 3 (n=366,343,356) | 83.6 [79.4 to 87.3] | 80.8 [76.2 to 84.8] | 88.5 [84.7 to 91.6]
  Additional serotypes - serotype 5 (n=368,343,357) | 99.7 [98.5 to 100.0] | 99.4 [97.9 to 99.9] | 99.7 [98.4 to 100.0]
  Additional serotypes - serotype 6A (n=366,342,355) | 100.0 [99.0 to 100.0] | 100.0 [98.9 to 100.0] | 99.7 [98.4 to 100.0]
  Additional serotypes - serotype 7F (n=366,343,358) | 100.0 [99.0 to 100.0] | 99.4 [97.9 to 99.9] | 99.4 [98.0 to 99.9]
  Additional serotype - serotype 19A (n=362,341,353) | 100.0 [99.0 to 100.0] | 100.0 [98.9 to 100.0] | 100.0 [99.0 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.1, 95% CI 2-sided [-1.61 to 1.81] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 2: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.8, 95% CI 2-sided [-2.39 to 0.23] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 3: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.9, 95% CI 2-sided [-2.54 to 0.20] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 4: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.02 to 1.11] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 5: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.03 to 1.04] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 6: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.13 to 1.06] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 7: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.25 to 1.37] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 8: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.6, 95% CI 2-sided [-0.76 to 2.18] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 9: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.5, 95% CI 2-sided [-0.87 to 2.18] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 10: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.3, 95% CI 2-sided [-0.74 to 1.62] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 11: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.03 to 1.04] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 12: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.3, 95% CI 2-sided [-1.61 to 0.76] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 13: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.4, 95% CI 2-sided [-1.52 to 2.39] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 14: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.5, 95% CI 2-sided [-2.30 to 1.04] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 15: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.9, 95% CI 2-sided [-2.87 to 0.74] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 16: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.5, 95% CI 2-sided [-2.55 to 1.50] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 17: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -1.1, 95% CI 2-sided [-3.06 to 0.57] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 18: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.6, 95% CI 2-sided [-2.44 to 1.00] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 19: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.3, 95% CI 2-sided [-1.21 to 2.05] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 20: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 1.1, 95% CI 2-sided [-0.52 to 3.16] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 21: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.8, 95% CI 2-sided [-1.05 to 2.87] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 22: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.9, 95% CI 2-sided [-0.17 to 2.53] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 23: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.8, 95% CI 2-sided [-0.20 to 2.44] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 24: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.0, 95% CI 2-sided [-1.79 to 1.66] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 25: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 2.8, 95% CI 2-sided [-2.85 to 8.55] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 26: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -4.9, 95% CI 2-sided [-9.99 to 0.21] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 27: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -7.7, 95% CI 2-sided [-13.14 to -2.37] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 28: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.3, 95% CI 2-sided [-1.00 to 1.84] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 29: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.27 to 1.30] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 30: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.3, 95% CI 2-sided [-1.84 to 1.02] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 31: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.04 to 1.08] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 32: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.3, 95% CI 2-sided [-0.76 to 1.56] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 33: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.3, 95% CI 2-sided [-0.83 to 1.56] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 34: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.6, 95% CI 2-sided [-0.47 to 2.09] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 35: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.6, 95% CI 2-sided [-0.48 to 2.00] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 36: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.0, 95% CI 2-sided [-1.59 to 1.49] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 37: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.04 to 1.09] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 38: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.05 to 1.04] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 39: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.09 to 1.07] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage

7. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥1.00 Mcg/mL in the Combined 13vPnC Group 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥1.00 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable immunogenicity population; (n)=number of subjects with a determinate IgG antibody concentration to the given serotype for the combined 13vPnC lot.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | Combined 13vPnC
Number analyzed (Participants) | 1213
observed percentage of participants
  Common serotypes - serotype 4 (n=1213) | 70.7 [68.1 to 73.3]
  Common serotypes - serotype 6B (n=1206) | 78.9 [76.4 to 81.1]
  Common serotypes - serotype 9V (n=1210) | 55.7 [52.9 to 58.5]
  Common serotypes - serotype 14 (n=1172) | 95.2 [93.8 to 96.4]
  Common serotypes - serotype 18C (n=1212) | 68.7 [66.0 to 71.3]
  Common serotypes - serotype 19F (n=1205) | 85.4 [83.3 to 87.3]
  Common serotypes - serotype 23F (n=1212) | 60.1 [57.2 to 62.8]
  Additional serotypes - serotype 1 (n=1209) | 75.2 [72.7 to 77.6]
  Additional serotypes - serotype 3 (n=1190) | 21.3 [19.0 to 23.8]
  Additional serotypes - serotype 5 (n=1207) | 60.3 [57.5 to 63.1]
  Additional serotypes - serotype 6A (n=1213) | 85.1 [82.9 to 87.0]
  Additional serotypes - serotype 7F (n=1210) | 92.8 [91.2 to 94.2]
  Additional serotypes - serotype 19A (n=1211) | 80.8 [78.4 to 82.9]

8. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥1.00 Mcg/mL in the Three 13vPnC Groups 1 Month After the Toddler Dose
Description: as for outcome 7
Time Frame: 1 month after the toddler dose (13 months of age)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot)
Number analyzed (Participants) | 415 | 397 | 408
observed percentage of participants
  Common serotypes - serotype 4 (n=364,342,355) | 86.0 [82.0 to 89.4] | 87.4 [83.4 to 90.7] | 92.7 [89.5 to 95.2]
  Common serotypes - serotype 6B (n=368,341,357) | 99.5 [98.1 to 99.9] | 99.1 [97.5 to 99.8] | 99.7 [98.4 to 100.0]
  Common serotypes - serotype 9V (n=368,342,357) | 80.7 [76.3 to 84.6] | 84.5 [80.2 to 88.2] | 85.4 [81.3 to 88.9]
  Common serotypes - serotype 14 (n=366,344,358) | 98.6 [96.8 to 99.6] | 98.8 [97.0 to 99.7] | 98.3 [96.4 to 99.4]
  Common serotypes - serotype 18C (n=362,341,354) | 79.6 [75.0 to 83.6] | 85.0 [80.8 to 88.7] | 89.5 [85.9 to 92.5]
  Common serotypes - serotype 19F (n=362,342,353) | 94.5 [91.6 to 96.6] | 95.3 [92.5 to 97.3] | 97.7 [95.6 to 99.0]
  Common serotypes - serotype 23F (n=362,340,353) | 91.7 [88.4 to 94.3] | 91.2 [87.6 to 94.0] | 89.8 [86.2 to 92.8]
  Additional serotypes - serotype 1 (n=367,344,357) | 91.8 [88.5 to 94.4] | 91.0 [87.5 to 93.8] | 94.4 [91.5 to 96.5]
  Additional serotypes - serotype 3 (n=366,343,356) | 32.0 [27.2 to 37.0] | 30.3 [25.5 to 35.5] | 36.8 [31.8 to 42.0]
  Additional serotypes - serotype 5 (n=368,343,357) | 94.0 [91.1 to 96.2] | 91.0 [87.4 to 93.8] | 93.6 [90.5 to 95.9]
  Additional serotypes - serotype 6A (n=366,342,355) | 99.2 [97.6 to 99.8] | 98.2 [96.2 to 99.4] | 99.2 [97.6 to 99.8]
  Additional serotypes - serotype 7F (n=366,343,358) | 98.1 [96.1 to 99.2] | 96.2 [93.6 to 98.0] | 98.6 [96.8 to 99.5]
  Additional serotype - serotype 19A (n=362,341,353) | 100.0 [99.0 to 100.0] | 99.4 [97.9 to 99.9] | 99.7 [98.4 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -1.4, 95% CI 2-sided [-6.52 to 3.63] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 2: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -6.7, 95% CI 2-sided [-11.30 to -2.15] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 3: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -5.2, 95% CI 2-sided [-9.85 to -0.79] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 4: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.3, 95% CI 2-sided [-1.19 to 2.07] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 5: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.3, 95% CI 2-sided [-1.69 to 1.06] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 6: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.6, 95% CI 2-sided [-2.27 to 0.75] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 7: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -3.8, 95% CI 2-sided [-9.46 to 1.82] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 8: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -4.7, 95% CI 2-sided [-10.24 to 0.76] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 9: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.9, 95% CI 2-sided [-6.30 to 4.41] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 10: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.2, 95% CI 2-sided [-2.14 to 1.73] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 11: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.3, 95% CI 2-sided [-1.69 to 2.39] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 12: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.5, 95% CI 2-sided [-1.46 to 2.59] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 13: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -5.5, 95% CI 2-sided [-11.17 to 0.20] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 14: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -10.0, 95% CI 2-sided [-15.31 to -4.70] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 15: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -4.5, 95% CI 2-sided [-9.55 to 0.46] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 16: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.8, 95% CI 2-sided [-4.23 to 2.52] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 17: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -3.3, 95% CI 2-sided [-6.35 to -0.40] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 18: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -2.4, 95% CI 2-sided [-5.44 to 0.33] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 19: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.5, 95% CI 2-sided [-3.67 to 4.80] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 20: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 1.9, 95% CI 2-sided [-2.38 to 6.28] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 21: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 1.4, 95% CI 2-sided [-3.06 to 5.82] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 22: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.8, 95% CI 2-sided [-3.34 to 5.08] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 23: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -2.6, 95% CI 2-sided [-6.39 to 1.18] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 24: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -3.4, 95% CI 2-sided [-7.45 to 0.46] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 25: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 1.6, 95% CI 2-sided [-5.20 to 8.55] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 26: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -4.8, 95% CI 2-sided [-11.79 to 2.16] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 27: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -6.5, 95% CI 2-sided [-13.51 to 0.54] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 28: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 3.1, 95% CI 2-sided [-0.84 to 7.13] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 29: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.5, 95% CI 2-sided [-3.14 to 4.11] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 30: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -2.6, 95% CI 2-sided [-6.72 to 1.40] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 31: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.9, 95% CI 2-sided [-0.87 to 3.02] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 32: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.0, 95% CI 2-sided [-1.62 to 1.71] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 33: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.9, 95% CI 2-sided [-3.00 to 0.92] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 34: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 1.9, 95% CI 2-sided [-0.62 to 4.67] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 35: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.5, 95% CI 2-sided [-2.67 to 1.55] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 36: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -2.4, 95% CI 2-sided [-5.11 to -0.01] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 37: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.6, 95% CI 2-sided [-0.45 to 2.10] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 38: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = 0.3, 95% CI 2-sided [-0.75 to 1.58] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage
Statistical Analysis 39: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Non-Inferiority or Equivalence — The equivalence test of Wiens and Iglewicz used to evaluate consistency among the three 13vPnC lots; Difference = -0.3, 95% CI 2-sided [-1.86 to 1.05] — Exact unconditional 2-sided 95% CI on the pairwise difference in proportions; expressed as a percentage

9. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody in the Three 13vPnC Groups 1 Month After the Toddler Dose
Description: Antibody geometric mean concentration (GMC) as measured by mcg/mL for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after the toddler dose (13 months of age)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: GMC mcg/mL
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot)
Number analyzed (Participants) | 415 | 397 | 408
GMC mcg/mL
  Common serotypes - serotype 4 (n=364,342,355) | 2.29 [2.11 to 2.48] | 2.25 [2.07 to 2.44] | 3.06 [2.79 to 3.35]
  Common serotypes - serotype 6B (n=368,341,357) | 11.14 [10.24 to 12.11] | 9.33 [8.55 to 10.19] | 9.92 [9.15 to 10.75]
  Common serotypes - serotype 9V (n=368,342,357) | 1.91 [1.76 to 2.06] | 1.95 [1.80 to 2.10] | 1.99 [1.84 to 2.15]
  Common serotypes - serotype 14 (n=366,344,358) | 6.61 [6.06 to 7.22] | 7.05 [6.42 to 7.74] | 6.91 [6.32 to 7.56]
  Common serotypes - serotype 18C (n=362,341,354) | 1.95 [1.78 to 2.12] | 2.20 [2.01 to 2.41] | 2.48 [2.27 to 2.71]
  Common serotypes - serotype 19F (n=362,342,353) | 4.51 [4.05 to 5.03] | 4.67 [4.23 to 5.14] | 6.51 [5.91 to 7.18]
  Common serotypes - serotype 23F (n=362,340,353) | 3.35 [3.02 to 3.71] | 3.46 [3.14 to 3.82] | 3.10 [2.81 to 3.43]
  Additional serotypes - serotype 1 (n=367,344,357) | 2.75 [2.53 to 2.99] | 2.95 [2.68 to 3.24] | 3.01 [2.75 to 3.30]
  Additional serotypes - serotype 3 (n=366,343,356) | 0.75 [0.69 to 0.81] | 0.71 [0.65 to 0.77] | 0.80 [0.74 to 0.87]
  Additional serotypes - serotype 5 (n=368,343,357) | 3.11 [2.87 to 3.37] | 2.63 [2.42 to 2.87] | 2.80 [2.60 to 3.02]
  Additional serotypes - serotype 6A (n=366,342,355) | 7.52 [6.93 to 8.17] | 6.97 [6.41 to 7.59] | 6.83 [6.30 to 7.41]
  Additional serotypes - serotype 7F (n=366,343,358) | 4.35 [4.01 to 4.72] | 4.24 [3.86 to 4.66] | 4.58 [4.21 to 4.98]
  Additional serotype - serotype 19A (n=362,341,353) | 8.41 [7.73 to 9.14] | 8.32 [7.66 to 9.04] | 8.60 [7.91 to 9.36]
Statistical Analysis 1: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 4; Test type: Superiority or Other; Difference in log-transformed GM = 0.02, 95% CI 2-sided [-0.10 to 0.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Superiority or Other; Difference in log-transformed GM = -0.29, 95% CI 2-sided [-0.41 to -0.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 4; Test type: Superiority or Other; Difference in log-transformed GM = -0.31, 95% CI 2-sided [-0.43 to -0.19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 6B; Test type: Superiority or Other; Difference in log-transformed GM = 0.18, 95% CI 2-sided [0.06 to 0.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Superiority or Other; Difference in log-transformed GM = 0.12, 95% CI 2-sided [-0.00 to 0.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 6B; Test type: Superiority or Other; Difference in log-transformed GM = -0.06, 95% CI 2-sided [-0.18 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 9V; Test type: Superiority or Other; Difference in log-transformed GM = -0.02, 95% CI 2-sided [-0.13 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Superiority or Other; Difference in log-transformed GM = -0.04, 95% CI 2-sided [-0.15 to 0.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 9V; Test type: Superiority or Other; Difference in log-transformed GM = -0.02, 95% CI 2-sided [-0.13 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 14; Test type: Superiority or Other; Difference in log-transformed GM = -0.06, 95% CI 2-sided [-0.19 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Superiority or Other; Difference in log-transformed GM = -0.04, 95% CI 2-sided [-0.17 to 0.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 14; Test type: Superiority or Other; Difference in log-transformed GM = 0.02, 95% CI 2-sided [-0.11 to 0.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 18C; Test type: Superiority or Other; Difference in log-transformed GM = -0.12, 95% CI 2-sided [-0.25 to 0.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Superiority or Other; Difference in log-transformed GM = -0.24, 95% CI 2-sided [-0.37 to -0.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 18C; Test type: Superiority or Other; Difference in log-transformed GM = -0.12, 95% CI 2-sided [-0.25 to 0.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 19F; Test type: Superiority or Other; Difference in log-transformed GM = -0.03, 95% CI 2-sided [-0.18 to 0.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Superiority or Other; Difference in log-transformed GM = -0.37, 95% CI 2-sided [-0.51 to -0.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 19F; Test type: Superiority or Other; Difference in log-transformed GM = -0.33, 95% CI 2-sided [-0.47 to -0.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Common serotypes - serotype 23F; Test type: Superiority or Other; Difference in log-transformed GM = -0.03, 95% CI 2-sided [-0.17 to 0.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Superiority or Other; Difference in log-transformed GM = 0.08, 95% CI 2-sided [-0.07 to 0.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Common serotypes - serotype 23F; Test type: Superiority or Other; Difference in log-transformed GM = 0.11, 95% CI 2-sided [-0.03 to 0.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 1; Test type: Superiority or Other; Difference in log-transformed GM = -0.07, 95% CI 2-sided [-0.20 to 0.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Superiority or Other; Difference in log-transformed GM = -0.09, 95% CI 2-sided [-0.21 to 0.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 1; Test type: Superiority or Other; Difference in log-transformed GM = -0.02, 95% CI 2-sided [-0.15 to 0.11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 3; Test type: Superiority or Other; Difference in log-transformed GM = 0.06, 95% CI 2-sided [-0.06 to 0.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Superiority or Other; Difference in log-transformed GM = -0.07, 95% CI 2-sided [-0.18 to 0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 3; Test type: Superiority or Other; Difference in log-transformed GM = -0.13, 95% CI 2-sided [-0.25 to -0.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 5; Test type: Superiority or Other; Difference in log-transformed GM = 0.17, 95% CI 2-sided [0.05 to 0.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 29: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Superiority or Other; Difference in log-transformed GM = 0.10, 95% CI 2-sided [-0.00 to 0.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 30: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 5; Test type: Superiority or Other; Difference in log-transformed GM = -0.06, 95% CI 2-sided [-0.17 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 31: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 6A; Test type: Superiority or Other; Difference in log-transformed GM = 0.08, 95% CI 2-sided [-0.04 to 0.19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 32: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Superiority or Other; Difference in log-transformed GM = 0.10, 95% CI 2-sided [-0.02 to 0.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 33: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 6A; Test type: Superiority or Other; Difference in log-transformed GM = 0.02, 95% CI 2-sided [-0.10 to 0.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 34: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 7F; Test type: Superiority or Other; Difference in log-transformed GM = 0.03, 95% CI 2-sided [-0.10 to 0.15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 35: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Superiority or Other; Difference in log-transformed GM = -0.05, 95% CI 2-sided [-0.17 to 0.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 36: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 7F; Test type: Superiority or Other; Difference in log-transformed GM = -0.08, 95% CI 2-sided [-0.20 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 37: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Pilot Lot 2); Additional serotypes - serotype 19A; Test type: Superiority or Other; Difference in log-transformed GM = 0.01, 95% CI 2-sided [-0.11 to 0.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 38: Comparison: 13vPnC (Pilot Lot 1) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Superiority or Other; Difference in log-transformed GM = -0.02, 95% CI 2-sided [-0.14 to 0.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 39: Comparison: 13vPnC (Pilot Lot 2) vs 13vPnC (Manufacturing Lot); Additional serotypes - serotype 19A; Test type: Superiority or Other; Difference in log-transformed GM = -0.03, 95% CI 2-sided [-0.15 to 0.08] — [estimate comment as in outcome 1, analysis 1]

10. Other Pre Specified Outcome: Percentage of Participants Reporting Local Reactions in the Three 13vPnC Groups and 7vPnC Group: Infant Series Dose 1 (2 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Induration and erythema were scaled as Any (induration or erythema present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 7 days after dose (2 months of age)
Population: Safety population: all participants who received at least 1 dose of study vaccine. N=number of participants reporting any local reactions; (n)=number of participants reporting yes for at least 1 day or no for all days for the three 13vPnC groups and 7vPnC, respectively.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC (Pilot Lot 1); 13vPnC (Pilot Lot 2); 13vPnC (Manufacturing Lot): Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 1 at 2, 4, and 6 months of age (Infant series Dose 1, 2, and 3, respectively); coadministered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age (infant series).
- 7vPnC: Participants received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) pilot lot 1 at 2, 4, and 6 months of age (Infant series Dose 1, 2, and 3, respectively); coadministered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age (infant series).
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Number analyzed (Participants) | 425 | 416 | 407 | 214
percentage of participants
  Tenderness: Any (n=420, 409, 400, 212) | 62.4 | 64.1 | 62.5 | 67.0
  Tenderness: Significant (n=348, 337, 345, 170) | 9.2 | 10.4 | 10.4 | 12.9
  Induration: Any (n=356, 347, 352, 176) | 16.6 | 19.6 | 19.3 | 18.2
  Induration: Mild (n=353, 344, 348, 173) | 14.7 | 16.9 | 15.5 | 16.2
  Induration: Moderate (n=338, 328, 340, 167) | 3.6 | 5.8 | 5.0 | 3.6
  Induration: Severe (n=333, 325, 335, 164) | 0.0 | 0.0 | 0.0 | 0.0
  Erythema: Any (n=355, 352, 360, 180) | 19.4 | 25.0 | 23.1 | 22.8
  Erythema: Mild (n=354, 352, 358, 180) | 18.1 | 24.7 | 21.2 | 21.7
  Erythema: Moderate (n=334, 326, 337, 164) | 2.1 | 0.6 | 2.4 | 1.2
  Erythema: Severe (n=333, 325, 335, 164) | 0.0 | 0.0 | 0.0 | 0.0

11. Other Pre Specified Outcome: Percentage of Participants Reporting Local Reactions in the Three 13vPnC Groups and 7vPnC Group: Infant Series Dose 2 (4 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Induration and erythema were scaled as Any (induration or erythema present); Mild (0.5 cm to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 7 days after dose (4 months of age)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Number analyzed (Participants) | 361 | 345 | 349 | 180
percentage of participants
  Tenderness: Any (n=354, 330, 337, 176) | 66.4 | 67.3 | 65.0 | 64.8
  Tenderness: Significant (n=269, 231, 262, 132) | 9.7 | 7.4 | 12.2 | 11.4
  Induration: Any (n=291, 248, 279, 141) | 24.4 | 22.6 | 28.7 | 17.7
  Induration: Mild (n=288, 246, 276, 141) | 22.6 | 22.0 | 26.8 | 17.7
  Induration: Moderate (n=270, 224, 255, 128) | 4.1 | 1.3 | 4.7 | 3.9
  Induration: Severe (n=263, 221, 250, 127) | 0.0 | 0.0 | 0.4 | 0.0
  Erythema: Any (n=292, 265, 281, 153) | 30.1 | 35.8 | 34.5 | 30.1
  Erythema: Mild (n=289, 263, 279, 153) | 28.4 | 34.6 | 33.3 | 28.8
  Erythema: Moderate (n=268, 223, 252, 128) | 3.4 | 1.8 | 3.2 | 3.1
  Erythema: Severe (n=263, 221, 249, 127) | 0.0 | 0.0 | 0.0 | 0.0

12. Other Pre Specified Outcome: Percentage of Participants Reporting Local Reactions in the Three 13vPnC Groups and 7vPnC Group: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 11
Time Frame: Within 7 days after dose (6 months of age)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Number analyzed (Participants) | 333 | 321 | 320 | 165
percentage of participants
  Tenderness: Any (n=317, 304, 300, 156) | 62.5 | 60.9 | 55.0 | 64.7
  Tenderness: Significant (n=248, 226, 237, 118) | 8.9 | 7.5 | 10.1 | 11.9
  Induration: Any (n=263, 250, 262, 128) | 27.0 | 23.6 | 28.6 | 30.5
  Induration: Mild (n=260, 249, 260, 127) | 24.6 | 22.5 | 27.3 | 29.1
  Induration: Moderate (n=242, 221, 229, 114) | 4.1 | 4.1 | 3.9 | 7.0
  Induration: Severe (n=237, 217, 227, 111) | 0.0 | 0.0 | 0.0 | 0.0
  Erythema: Any (n=278, 262, 274, 137) | 39.6 | 35.9 | 37.6 | 39.4
  Erythema: Mild (n=275, 260, 272, 135) | 37.1 | 33.8 | 36.4 | 38.5
  Erythema: Moderate (n=243, 219, 231, 116) | 5.3 | 4.1 | 5.6 | 7.8
  Erythema: Severe (n=237, 217, 227, 111) | 0.0 | 0.0 | 0.0 | 0.0

13. Other Pre Specified Outcome: Percentage of Participants Reporting Local Reactions in the Combined 13vPnC Group and 7vPnC Group: Toddler Dose (12 Months of Age)
Description: as for outcome 11
Time Frame: Within 7 days after dose (12 months of age)
Population: Safety population: all participants who received at least 1 dose of study vaccine. N=number of participants reporting any local reactions; (n)=number of participants reporting yes for at least 1 day or no for all days for the combined 13vPnC group and 7vPnC, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Combined 13vPnC | 7vPnC
Number analyzed (Participants) | 889 | 106
percentage of participants
  Tenderness: Any (n=826, 131) | 57.3 | 63.4
  Tenderness: Significant (n=630, 97) | 6.7 | 4.1
  Induration: Any (n=698, 110) | 31.5 | 43.6
  Induration: Mild (n=689, 107) | 28.9 | 41.1
  Induration: Moderate (n=627, 101) | 8.5 | 17.8
  Induration: Severe (n=603, 93) | 0.0 | 0.0
  Erythema: Any (n=749, 121) | 42.6 | 52.9
  Erythema: Mild (n=735, 116) | 39.2 | 50.0
  Erythema: Moderate (n=631, 104) | 10.6 | 21.2
  Erythema: Severe (n=603, 93) | 0.0 | 0.0

14. Other Pre Specified Outcome: Percentage of Participants Reporting Systemic Events in the Three 13vPnC Groups and 7vPnC Group: Infant Series Dose 1 (2 Months of Age)
Description: Systemic events (any fever ≥ 38 degrees Celsius [C], decreased appetite, irritability, increased sleep, decreased sleep, and hives [urticaria]) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after dose (2 months of age)
Population: Safety population: all participants who received at least 1 dose of study vaccine. N=number of participants reporting any systemic events; (n)=number of participants reporting yes for at least 1 day or no for all days for the three 13vPnC groups and 7vPnC, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Number analyzed (Participants) | 465 | 457 | 456 | 237
percentage of participants
  Fever ≥38 but ≤39 degrees C (n=353, 337, 353, 173) | 24.6 | 23.4 | 24.6 | 26.0
  Fever >39 but ≤40 degrees C (n=328, 319, 333, 161) | 0.6 | 0.3 | 0.9 | 1.2
  Fever >40 degrees C (n=328, 319, 331, 160) | 0.0 | 0.0 | 0.3 | 0.6
  Decreased appetite (n=393, 385, 386, 200) | 50.6 | 46.0 | 50.0 | 49.0
  Irritability (n=435, 432, 433, 226) | 85.7 | 84.3 | 89.1 | 87.6
  Increased sleep (n=425, 417, 402, 212) | 71.5 | 72.7 | 69.4 | 72.6
  Decreased sleep (n=379, 377, 377, 194) | 44.1 | 46.9 | 42.2 | 46.4
  Hives [urticaria] (n=333, 328, 335, 164) | 0.6 | 0.9 | 0.6 | 0.0

15. Other Pre Specified Outcome: Percentage of Participants Reporting Systemic Events in the Three 13vPnC Groups and 7vPnC Group: Infant Series Dose 2 (4 Months of Age)
Description: Systemic events (any fever ≥ 38 degrees C, decreased appetite, irritability, increased sleep, decreased sleep, and hives [urticaria]) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 7 days after dose (4 months of age)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Number analyzed (Participants) | 400 | 398 | 410 | 208
percentage of participants
  Fever ≥38 but ≤39 degrees C (n=290, 250, 290, 143) | 33.4 | 36.4 | 35.5 | 28.0
  Fever >39 but ≤40 degrees C (n=263, 216, 248, 124) | 3.4 | 3.2 | 3.6 | 0.0
  Fever >40 degrees C (n=259, 214, 245, 124) | 0.4 | 0.0 | 0.0 | 0.0
  Decreased appetite (n=322, 293, 325, 164) | 48.4 | 49.1 | 48.0 | 49.4
  Irritability (n=377, 370, 376, 201) | 86.5 | 86.5 | 84.6 | 81.1
  Increased sleep (n=332, 318, 343, 177) | 64.8 | 68.2 | 67.3 | 63.3
  Decreased sleep (n=324, 291, 305, 159) | 49.1 | 48.8 | 44.6 | 48.4
  Hives [urticaria] (n=263, 225, 253, 127) | 0.4 | 2.2 | 1.6 | 0.8

16. Other Pre Specified Outcome: Percentage of Participants Reporting Systemic Events in the Three 13vPnC Groups and 7vPnC Group: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 15
Time Frame: Within 7 days after dose (6 months of age)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC (Pilot Lot 1) | 13vPnC (Pilot Lot 2) | 13vPnC (Manufacturing Lot) | 7vPnC
Number analyzed (Participants) | 373 | 365 | 373 | 192
percentage of participants
  Fever ≥38 but ≤39 degrees C (n=266, 246, 252, 132) | 26.3 | 27.6 | 31.7 | 32.6
  Fever >39 but ≤40 degrees C (n=237, 219, 231, 113) | 2.5 | 3.7 | 5.6 | 6.2
  Fever >40 degrees C (n=234, 216, 224, 111) | 0.0 | 0.5 | 0.0 | 0.9
  Decreased appetite (n=286, 273, 286, 144) | 45.8 | 48.0 | 50.7 | 50.0
  Irritability (n=352, 339, 347, 186) | 79.5 | 80.5 | 82.7 | 84.4
  Increased sleep (n=289, 289, 286, 138) | 55.4 | 58.8 | 59.8 | 51.4
  Decreased sleep (n=282, 272, 289, 147) | 42.6 | 50.4 | 48.4 | 56.5
  Hives [urticaria] (n=239, 218, 229, 112) | 1.7 | 0.9 | 1.7 | 1.8

17. Other Pre Specified Outcome: Percentage of Participants Reporting Systemic Events in the Combined 13vPnC Group and 7vPnC Group: Toddler Dose (12 Months of Age)
Description: as for outcome 15
Time Frame: Within 7 days after dose (12 months of age)
Population: Safety population: all participants who received at least 1 dose of study vaccine. N=number of participants reporting any systemic events; (n)=number of participants reporting yes for at least 1 day or no for all days for the combined 13vPnC group and 7vPnC, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Combined 13vPnC | 7vPnC
Number analyzed (Participants) | 1001 | 171
percentage of participants
  Fever ≥38 but ≤39 degrees C (n=667, 107) | 28.8 | 29.9
  Fever >39 but ≤40 degrees C (n=592, 95) | 4.4 | 5.3
  Fever >40 degrees C (n=586, 93) | 1.0 | 0.0
  Decreased appetite (n=790, 115) | 51.9 | 50.4
  Irritability (n=943, 160) | 81.8 | 80.0
  Increased sleep (n=779, 126) | 47.8 | 47.6
  Decreased sleep (n=770, 117) | 46.9 | 42.7
  Hives [urticaria] (n=607, 96) | 2.1 | 5.2

ADVERSE EVENTS:
Time Frame: Baseline through 6 Month Follow-up after last study vaccination (18 Months). Local reactions and systemic events assessed within 7 days of dose: Infant Series Dose 1, 2, and 3 at 2, 4, and 6 months of age, respectively; Toddler Dose at 12 months of age.
Description: Safety population = all randomized subjects with at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Groups:
- Infant Series 13vPnC (Pilot Lot 1): Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 1 at 2, 4, and 6 months of age (infant series); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age (infant series).
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=407; systematic (solicited) Local Reactions N=262; systematic (solicited) Systemic Events N=373.
- Infant Series 13vPnC (Pilot Lot 2): Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 2 at 2, 4, and 6 months of age (infant series); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age (infant series).
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=394; systematic (solicited) Local Reactions N=262; systematic (solicited) Systemic Events N=364.
- Infant Series 13vPnC (Manufacturing Lot): Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) manufacturing lot (manu lot) at 2, 4, and 6 months of age (infant series); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age (infant series).
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=402; systematic (solicited) Local Reactions N=250; systematic (solicited) Systemic Events N=386.
- Infant Series 7vPnC: Participants received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 2, 4, and 6 months of age (infant series); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age (infant series).
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=207; systematic (solicited) Local Reactions N=142; systematic (solicited) Systemic Events N=198.
- After the Infant Series Combined 13vPnC: Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 1, 2, or manufacturing lot at 2, 4, and 6 months of age (assessment at 7 months of age; 1 month after the infant series); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age(assessment at 7 months of age; 1 month after the infant series).
- After the Infant Series 7vPnC: Participants received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 2, 4, and 6 months of age (assessment at 7 months of age; 1 month after the infant series); co-administered with Pediarix® (a commercially available combination diphtheria and tetanus toxoid; acellular pertussis and hepatitis B antigens; and inactivated poliovirus); and a commercially available Haemophilus influenzae type b (Hib) vaccine at 2, 4, and 6 months of age(assessment at 7 months of age; 1 month after the infant series).
- Toddler Dose Combined 13vPnC: Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 1, 2, or manufacturing lot at 12 months of age; co-administered with a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age.
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=434; systematic (solicited) Local Reactions N=473; systematic (solicited) Systemic Events N=771.
- Toddler Dose 7vPnC: Participants received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 12 months of age; co-administered with a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age.
  Other Adverse Events (non-serious events): the number affected (N) for non-systematic (unsolicited) Other Adverse Events N=75; systematic (solicited) Local Reactions N=83; systematic (solicited) Systemic Events N=128.
- Post Toddler Dose 6-Month Follow-up Combined 13vPnC: Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) pilot lot 1, 2, or manufacturing lot at 12 months of age (assessment at 18 months of age; 6 months after the toddler dose) ; co-administered with a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age (assessment at 18 months of age; 6 months after the toddler dose).
- Post Toddler Dose 6-Month Follow-up 7vPnC: Participants received 1 single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) at 12 months of age (assessment at 18 months of age; 6 months after the toddler dose) ; co-administered with a commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella), or if not available, a commercially available MMR and a commercially available varicella vaccine administered in separate injections; and a commercially available hepatitis A vaccine (HAV) administered at 12 months of age (assessment at 18 months of age; 6 months after the toddler dose).
Arm/Group | Infant Series 13vPnC (Pilot Lot 1) | Infant Series 13vPnC (Pilot Lot 2) | Infant Series 13vPnC (Manufacturing Lot) | Infant Series 7vPnC | After the Infant Series Combined 13vPnC | After the Infant Series 7vPnC | Toddler Dose Combined 13vPnC | Toddler Dose 7vPnC | Post Toddler Dose 6-Month Follow-up Combined 13vPnC | Post Toddler Dose 6-Month Follow-up 7vPnC
Serious Adverse Events (participants affected / at risk) | 13/486 | 23/483 | 17/483 | 15/244 | 25/1445 | 3/244 | 9/1210 | 1/208 | 21/1443 | 7/244
Other Adverse Events (participants affected / at risk) | 407/486 | 394/483 | 402/483 | 207/244 | 88/1445 | 11/244 | 771/1210 | 128/208 | 37/1443 | 9/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant Series 13vPnC (Pilot Lot 1) (N=486) | Infant Series 13vPnC (Pilot Lot 2) (N=483) | Infant Series 13vPnC (Manufacturing Lot) (N=483) | Infant Series 7vPnC (N=244) | After the Infant Series Combined 13vPnC (N=1445) | After the Infant Series 7vPnC (N=244) | Toddler Dose Combined 13vPnC (N=1210) | Toddler Dose 7vPnC (N=208) | Post Toddler Dose 6-Month Follow-up Combined 13vPnC (N=1443) | Post Toddler Dose 6-Month Follow-up 7vPnC (N=244)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Sudden infant death syndrome (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergy to vaccine (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 5 | 2 | 4 | 2 | 2 | 0 | 0 | 1 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 5 | 4 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 3 | 1
Respiratory syncytial virus infection (Infections and infestations) | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 1
Otitis media (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abscess oral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis enteroviral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0
Eczema herpeticum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis pharyngeal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infant Series 13vPnC (Pilot Lot 1) (N=486) | Infant Series 13vPnC (Pilot Lot 2) (N=483) | Infant Series 13vPnC (Manufacturing Lot) (N=483) | Infant Series 7vPnC (N=244) | After the Infant Series Combined 13vPnC (N=1445) | After the Infant Series 7vPnC (N=244) | Toddler Dose Combined 13vPnC (N=1210) | Toddler Dose 7vPnC (N=208) | Post Toddler Dose 6-Month Follow-up Combined 13vPnC (N=1443) | Post Toddler Dose 6-Month Follow-up 7vPnC (N=244)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 4 | 0 | 2 | 0 | 4 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 9 | 6 | 11 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macrocephaly (Congenital, familial and genetic disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brachycephaly (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemihypertrophy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypospadias (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngomalacia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Naevus flammeus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary valve stenosis congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skull malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Von Willebrand's disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Congenital neavus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tibial torsion (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 6 | 7 | 6 | 8 | 0 | 0 | 4 | 1 | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 1 | 2 | 4 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Precocious puberty (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 35 | 37 | 44 | 26 | 0 | 1 | 17 | 3 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 3 | 3 | 2 | 4 | 1 | 0 | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 4 | 5 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dark circles under eyes (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heterophoria (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pupillary reflex impaired (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scleral disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 44 | 34 | 56 | 32 | 1 | 0 | 37 | 8 | 0 | 0
Vomiting (Gastrointestinal disorders) | 26 | 23 | 30 | 25 | 0 | 0 | 17 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 15 | 31 | 17 | 17 | 1 | 1 | 3 | 3 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 28 | 20 | 18 | 10 | 2 | 0 | 3 | 0 | 0 | 1
Teething (Gastrointestinal disorders) | 5 | 11 | 9 | 2 | 0 | 0 | 7 | 1 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 3 | 5 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 6 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 3 | 0 | 5 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingval cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingval ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue geographic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting projectile (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Anal skin tags (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 43 | 49 | 40 | 25 | 0 | 0 | 38 | 9 | 0 | 0
Irritability (General disorders) | 15 | 12 | 7 | 8 | 0 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 4 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Injection site swelling (General disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Injection site induration (General disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Injection site reaction (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site dryness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Developmental delay (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 2 | 2 | 4 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 4 | 0 | 3 | 0 | 6 | 0
Food allergy (Immune system disorders) | 0 | 1 | 1 | 0 | 4 | 1 | 4 | 0 | 3 | 1
Allergy to vaccine (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 194 | 187 | 204 | 97 | 2 | 0 | 62 | 11 | 0 | 1
Otitis media (Infections and infestations) | 142 | 125 | 135 | 85 | 4 | 0 | 70 | 20 | 1 | 1
Bronchiolitis (Infections and infestations) | 72 | 75 | 66 | 44 | 1 | 0 | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 31 | 29 | 28 | 17 | 0 | 0 | 12 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 21 | 32 | 19 | 15 | 1 | 0 | 16 | 3 | 0 | 0
Viral infection (Infections and infestations) | 19 | 18 | 24 | 11 | 0 | 0 | 20 | 6 | 0 | 0
Croup infectious (Infections and infestations) | 16 | 19 | 18 | 8 | 0 | 0 | 10 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 21 | 14 | 10 | 7 | 0 | 0 | 2 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 16 | 15 | 11 | 10 | 0 | 0 | 12 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 14 | 14 | 15 | 6 | 0 | 0 | 8 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 11 | 16 | 13 | 6 | 1 | 0 | 11 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 11 | 10 | 12 | 7 | 0 | 1 | 11 | 4 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 8 | 6 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 7 | 7 | 10 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 9 | 12 | 4 | 8 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 6 | 12 | 2 | 0 | 0 | 3 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 11 | 11 | 7 | 2 | 0 | 0 | 3 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 10 | 5 | 9 | 5 | 0 | 0 | 2 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 5 | 10 | 3 | 1 | 0 | 2 | 0 | 0 | 0
Candida nappy rash (Infections and infestations) | 7 | 5 | 9 | 3 | 0 | 0 | 2 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 9 | 5 | 6 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 5 | 5 | 7 | 4 | 0 | 0 | 5 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 4 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Viral skin infection (Infections and infestations) | 3 | 7 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 6 | 6 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Impetigo (Infections and infestations) | 2 | 2 | 2 | 3 | 0 | 0 | 3 | 0 | 0 | 0
Skin candida (Infections and infestations) | 1 | 4 | 3 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 2 | 2 | 2 | 1 | 0 | 0 | 5 | 0 | 0 | 0
Roseola (Infections and infestations) | 0 | 4 | 2 | 1 | 0 | 0 | 4 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 2 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0
Dacryocystitis (Infections and infestations) | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo candida (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatophytosis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema herpeticum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema infectiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scarlet fever (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 1 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0/1433 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Torus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 2 | 2 | 1 | 1 | 0 | 6 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur functional (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head circumference abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lead increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Body height below normal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 5 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 3 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeding disorder neonatal (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cow's milk intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overweight (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Head deformity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Muscle twiching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign penile neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Head titubation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural effusion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral cyst (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Speech disorder developmental (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gross motor delay (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Crying (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Screaming (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tic (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Penile adhesion (Reproductive system and breast disorders) | 1 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital labial adhesions (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 52 | 51 | 33 | 0 | 1 | 22 | 8 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 43 | 48 | 34 | 15 | 0 | 1 | 5 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 21 | 25 | 18 | 9 | 1 | 0 | 22 | 5 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 18 | 10 | 15 | 5 | 3 | 0 | 3 | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 8 | 6 | 6 | 2 | 1 | 0 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 1 | 4 | 0 | 3 | 1 | 10 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 1 | 10 | 2 | 4 | 1 | 4 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0/483 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 45 | 28 | 42 | 21 | 12 | 1 | 17 | 0 | 6 | 4
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 34 | 13 | 30 | 13 | 0 | 1 | 31 | 5 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 22 | 20 | 18 | 13 | 3 | 0 | 27 | 2 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 12 | 12 | 11 | 12 | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 9 | 12 | 15 | 9 | 4 | 0 | 4 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 11 | 8 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 4 | 9 | 4 | 1 | 0 | 1 | 1 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 7 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 8 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 8 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 3 | 5 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 2 | 2 | 6 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 4 | 2 | 1 | 0 | 0 | 6 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne infantile (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acanthosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Dermographism (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acrodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overfeeding of infant (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (any) (Skin and subcutaneous tissue disorders) | 262/420 | 262/409 | 250/400 | 142/212 | 0/0 | 0/0 | 473/826 | 83/131 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 235/354 | 222/330 | 219/337 | 114/176 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)=present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 198/317 | 185/304 | 165/300 | 101/156 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)=present at site of vaccination.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 32/348 | 35/337 | 36/345 | 22/170 | 0/0 | 0/0 | 42/630 | 4/97 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 26/269 | 17/231 | 32/262 | 15/132 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)=present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 22/248 | 17/226 | 24/237 | 14/118 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)=present and interfered with limb movement.
Induration (any) (Skin and subcutaneous tissue disorders) | 59/356 | 68/347 | 68/352 | 32/176 | 0/0 | 0/0 | 220/698 | 48/110 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (any)=present at site of vaccination.
Induration (any) (Skin and subcutaneous tissue disorders) | 71/291 | 56/248 | 80/279 | 25/141 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)=present at site of vaccination.
Induration (any) (Skin and subcutaneous tissue disorders) | 71/263 | 59/250 | 75/262 | 39/128 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (any)=present at site of vaccination.
Induration (mild) (Skin and subcutaneous tissue disorders) | 52/353 | 58/344 | 54/348 | 28/173 | 0/0 | 0/0 | 199/689 | 44/107 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (mild) (Skin and subcutaneous tissue disorders) | 65/288 | 54/246 | 74/276 | 25/141 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild)=0.5 cm to 2.0 cm.
Induration (mild) (Skin and subcutaneous tissue disorders) | 64/260 | 56/249 | 71/260 | 37/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild)=0.5 cm to 2.0 cm.
Induration (moderate) (Skin and subcutaneous tissue disorders) | 12/338 | 19/328 | 17/340 | 6/167 | 0/0 | 0/0 | 53/627 | 18/101 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (moderate) (Skin and subcutaneous tissue disorders) | 11/270 | 3/224 | 12/255 | 5/128 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (moderate) (Skin and subcutaneous tissue disorders) | 10/242 | 9/221 | 9/229 | 8/114 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/333 | 0/325 | 0/335 | 0/164 | 0/0 | 0/0 | 0/603 | 0/93 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/263 | 0/221 | 1/250 | 0/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe) >7.0 cm.
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/237 | 0/217 | 0/227 | 0/111 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe) >7.0 cm.
Erythema (any) (Skin and subcutaneous tissue disorders) | 69/355 | 88/352 | 83/360 | 41/180 | 0/0 | 0/0 | 319/749 | 64/121 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (any)=present at site of vaccination.
Erythema (any) (Skin and subcutaneous tissue disorders) | 88/292 | 95/265 | 97/281 | 46/153 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any)=present at site of vaccination.
Erythema (any) (Skin and subcutaneous tissue disorders) | 110/278 | 94/262 | 103/274 | 54/137 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (any)=present at site of vaccination.
Erythema (mild) (Skin and subcutaneous tissue disorders) | 64/354 | 87/352 | 76/358 | 39/180 | 0/0 | 0/0 | 288/735 | 58/116 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (mild) (Skin and subcutaneous tissue disorders) | 82/289 | 91/263 | 93/279 | 44/153 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (mild) (Skin and subcutaneous tissue disorders) | 102/275 | 88/260 | 99/272 | 52/135 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 7/334 | 2/326 | 8/337 | 2/164 | 0/0 | 0/0 | 67/631 | 22/104 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 9/268 | 4/223 | 8/252 | 4/128 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate)=2.5 cm to 7.0 cm
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 13/243 | 9/219 | 13/231 | 9/116 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/333 | 0/325 | 0/335 | 0/164 | 0/0 | 0/0 | 0/603 | 0/93 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/263 | 0/221 | 0/249 | 0/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe) >7.0 cm.
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/237 | 0/217 | 0/227 | 0/111 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (severe) >7.0 cm.
Fever ≥ 38 degrees Celsius C but ≤ 39 degrees C (General disorders) | 87/353 | 79/337 | 87/353 | 45/173 | 0/0 | 0/0 | 192/667 | 32/107 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥ 38 degrees Celsius C but ≤ 39 degrees C.
Fever ≥ 38 degrees Celsius C but ≤ 39 degrees C (General disorders) | 97/290 | 91/250 | 103/290 | 40/143 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥ 38 degrees Celsius C but ≤ 39 degrees C.
Fever ≥ 38 degrees Celsius C but ≤ 39 degrees C (General disorders) | 70/266 | 68/246 | 80/252 | 43/132 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥ 38 degrees Celsius C but ≤ 39 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 2/328 | 1/319 | 3/333 | 2/161 | 0/0 | 0/0 | 26/592 | 5/95 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever > 39 degrees C but ≤ 40 degrees C.
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 9/263 | 7/216 | 9/248 | 0/124 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 39 degrees C but ≤ 40 degrees C.
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 6/237 | 8/219 | 13/231 | 7/113 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 39 degrees C but ≤ 40 degrees C.
Fever > 40 degrees C (General disorders) | 0/328 | 0/319 | 1/331 | 1/160 | 0/0 | 0/0 | 6/586 | 0/93 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever > 40 degrees C.
Fever > 40 degrees C (General disorders) | 1/259 | 0/214 | 0/245 | 0/124 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 40 degrees C.
Fever > 40 degrees C (General disorders) | 0/234 | 1/216 | 0/224 | 1/111 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 40 degrees C.
Decreased appetite (General disorders) | 199/393 | 177/385 | 193/386 | 98/200 | 0/0 | 0/0 | 410/790 | 58/115 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite.
Decreased appetite (General disorders) | 156/322 | 144/293 | 156/325 | 81/164 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite.
Decreased appetite (General disorders) | 131/286 | 131/273 | 145/286 | 72/144 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite.
Irritability (General disorders) | 373/435 | 364/432 | 386/433 | 198/226 | 0/0 | 0/0 | 771/943 | 128/160 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability.
Irritability (General disorders) | 326/377 | 320/370 | 318/376 | 163/201 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability.
Irritability (General disorders) | 280/352 | 273/339 | 287/347 | 157/186 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability.
Increased sleep (General disorders) | 304/425 | 303/417 | 279/402 | 154/212 | 0/0 | 0/0 | 372/779 | 60/126 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep.
Increased sleep (General disorders) | 215/332 | 217/318 | 231/343 | 112/177 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep.
Increased sleep (General disorders) | 160/289 | 170/289 | 171/286 | 71/138 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep.
Decreased sleep (General disorders) | 167/379 | 177/377 | 159/377 | 90/194 | 0/0 | 0/0 | 361/770 | 50/117 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep.
Decreased sleep (General disorders) | 159/324 | 142/291 | 136/305 | 77/159 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep.
Decreased sleep (General disorders) | 120/282 | 137/272 | 140/289 | 83/147 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep.
Hives (Urticaria) (General disorders) | 2/333 | 3/328 | 2/335 | 0/164 | 0/0 | 0/0 | 13/607 | 5/96 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Hives (Urticaria).
Hives (Urticaria) (General disorders) | 1/263 | 5/225 | 4/253 | 1/127 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Hives (Urticaria).
Hives (Urticaria) (General disorders) | 4/239 | 2/218 | 4/229 | 2/112 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Hives (Urticaria).

LIMITATIONS AND CAVEATS:
Commercially available Measles, Mumps, and Rubella-varicella vaccine (MMR-varicella) was not available as planned; the alternate of a commercially available MMR and a commercially available varicella vaccine was administered in separate injections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.